CLINICAL TRIAL: NCT07257484
Title: Tirzepatide's Role in Postmenopausal HR+ Breast Cancer Survivors
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-06029016; KL2TR002385 (NIH)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Obesity (Disorder); Breast Cancer
Keywords: tirzepatide; hormone receptor positive; HR+; postmenopausal
MeSH Terms: conditions — Obesity; Breast Neoplasms | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug (Experimental)
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Participants will take tirzepatide weekly for 24 weeks. The dose will be adjusted on a monthly basis as clinically indicated.

SUMMARY:
This study will explore whether tirzepatide is a practical and acceptable treatment for postmenopausal women with a history of hormone receptor-positive breast cancer and obesity. The investigators aim to understand whether participants are willing and able to take this medication once weekly for 6 months and whether it may help improve weight and overall health. There will be monthly check-ins to monitor progress and safety. At the beginning and end of the study, participants will undergo body composition assessments, blood tests and a stool sample will be collected, and surveys will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female
* Age ≥ 18
* Obesity as defined by current BMI ≥ 30 kg/m²
* Postmenopausal as defined by one or more of the following

  * Age ≥60 years
  * Age <60 years with amenorrhea for ≥ 1 year
  * Documented bilateral surgical oophorectomy
  * Chemical menopause with the addition of LHRH agonists at least 12 weeks prior to enrolment, and plan to remain on LHRH agonists throughout the trial
* HR+ (ER and/or PR) stage 0-III breast cancer
* Completed curative treatment (surgery, chemotherapy, radiotherapy) at least 12 weeks prior to enrolment
* On adjuvant hormonal therapy (aromatase inhibitor or tamoxifen)
* Insurance approval for tirzepatide or willing to pay out of pocket
* Willing to provide informed consent and comply with study procedures

Exclusion Criteria:

* Stage IV breast cancer
* Concomitant use of CDK inhibitors
* Concomitant use of antiHER2 therapy
* The PI may be consulted regarding enrollment of women receiving other endocrine therapy medications
* Other active malignancy requiring treatment
* Enrollment in another investigational clinical trial
* Contraindication to tirzepatide
* Treatment with a GLP-1 receptor agonist within the last 3 months
* Diabetes requiring insulin
* Any disorder, unwillingness, or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardize the subject's safety or compliance with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-07-06 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants completing week 24 visit with all required assessments | 24 weeks

SECONDARY OUTCOMES:
Percent change in body weight from baseline to week 24 | Baseline, 24 weeks
Absolute change in visceral fat mass from baseline to week 24 | Baseline, 24 weeks
  As assessed by SECA scan
Percent change in visceral fat mass from baseline to week 24 | Baseline, 24 weeks
  As assessed by SECA scan
Absolute change in fasting glucose from baseline to week 24 | Baseline, 24 weeks
Percent change in fasting glucose from baseline to week 24 | Baseline, 24 weeks
Absolute change in fasting insulin from baseline to week 24 | Baseline, 24 weeks
Percent change in fasting insulin from baseline to week 24 | Baseline, 24 weeks
Absolute change in hemoglobin A1c from baseline to week 24 | Baseline, 24 weeks
Percent change in hemoglobin A1c from baseline to week 24 | Baseline, 24 weeks
Absolute change in IGF-1 from baseline to week 24 | Baseline, 24 weeks
Percent change in IGF-1 from baseline to week 24 | Baseline, 24 weeks
Absolute change in leptin from baseline to week 24 | Baseline, 24 weeks
Percent change in leptin from baseline to week 24 | Baseline, 24 weeks
Absolute change in adiponectin from baseline to week 24 | Baseline, 24 weeks
Percent change in adiponectin from baseline to week 24 | Baseline, 24 weeks
Absolute change in hs-CRP from baseline to week 24 | Baseline, 24 weeks
Percent change in hs-CRP from baseline to week 24 | Baseline, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Schmitz, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No